CLINICAL TRIAL: NCT06712888
Title: Toripalimab Versus Placebo Combined with Induction Chemotherapy Followed by Concurrent Chemoradiotherapy for Locoregionally Advanced Nasopharyngeal Carcinoma: a Multicenter, Randomized, Placebo-controlled, Double-blind, Phase 3 Trial
Brief Title: Toripalimab Vs. Placebo Wtih GP Induction Chemotherapy in Locoregionally Advanced Nasopharyngeal Carcinoma
Acronym: Navigation
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital of Guangxi Medical University (Other); Guangxi Medical University Cancer Center (Unknown); Affiliated Hospital of Guangdong Medical University (Other); Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other); The University of Hong Kong-Shenzhen Hospital (Other); Hunan Cancer Hospital (Other); The Affiliated Cancer Hosipital of Guizhou Meidical University (Unknown); Sichuan Cancer Hospital and Research Institute (Other); Fujian Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-FXY-323
Record Dates: First submitted 2024-11-25; First posted 2024-12-02 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
Keywords: Nasopharyngeal Carcinoma; Anti-PD-1 therapy; induction chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — toripalimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Induction GP+placebo group (Active Comparator): GP + Placebo Induction Therapy:
  Gemcitabine: 1000 mg/m² on days 1 and 8 DDP (cisplatin): 80 mg/m² on day 1 Placebo: 240 mg on day 1 Total of 3 cycles.
  Concurrent Chemoradiotherapy (CCRT):
  DDP (cisplatin): 100 mg/m² on day 1 of radiation, then every 3 weeks during radiotherapy.
  Total of 3 cycles (administered on D1, D22, and D43).
  Adjuvant Metronomic Capecitabine Therapy:
  Starts 4-6 weeks after the completion of radiotherapy and continues for up to 1 year.
  Adjuvant metronomi capecitabine is administered at the physician's discretion: Capecitabine: 650 mg/m², administered BID (twice daily).
  Interventions: Drug: GP plus placebo induction therapy
- Induction GP+toripalimab group (Experimental): Induction GP + Toripalimab Therapy:
  Gemcitabine: 1000 mg/m² on days 1 and 8 DDP (cisplatin): 80 mg/m² on day 1 Toripalimab: 240 mg on day 1 Total of 3 cycles.
  Concurrent Chemoradiotherapy (CCRT):
  DDP (cisplatin): 100 mg/m² on day 1 of radiation, then every 3 weeks during radiotherapy.
  Total of 3 cycles (administered on D1, D22, and D43).
  Adjuvant Metronomic Capecitabine Therapy:
  Starts 4-6 weeks after the completion of radiotherapy and continues for up to 1 year.
  Adjuvant metronomic capecitabine therapy is administered at the physician's discretion: Capecitabine: 650 mg/m², administered BID (twice daily).
  Interventions: Drug: TORIPALIMAB INJECTION (JS001 ) combine with GP chemotherapy

INTERVENTIONS:
Drug: TORIPALIMAB INJECTION (JS001 ) combine with GP chemotherapy — Drug: Toripalimab 240mg will be given every 3 weeks for 3 cycles, started on day 1 of induction chemotherapy.
  Other Names:
  JS001 PD-1 antibody
  Drug: Gemcitabine 1000mg/m2, d1 & 8 of every cycle, every 3 weeks for 3 cycles before radiation.
  Drug: Cisplatin Induction cisplatin 80mg/m2, every 3 weeks for 3 cycles before radiation; Concurrent cisplatin 100mg/m2, every 3 weeks for 3 cycles during radiation
  Other Names:
  DDP
  Radiation: intensity-modulated radiotherapy Definitive intensity-modulated radiotherapy (IMRT) of 70 Gy will be given in 33 fractions.
  Other Names:
  IMRT
  Arms: Induction GP+toripalimab group
Drug: GP plus placebo induction therapy — Drug: Placebo 240mg will be given every 3 weeks for 3 cycles, started on day 1 of induction chemotherapy.
  Drug: Gemcitabine 1000mg/m2, d1 & 8 of every cycle, every 3 weeks for 3 cycles before radiation.
  Drug: Cisplatin Induction cisplatin 80mg/m2, every 3 weeks for 3 cycles before radiation; Concurrent cisplatin 100mg/m2, every 3 weeks for 3 cycles during radiation
  Other Names:
  DDP Radiation: intensity-modulated radiotherapy Definitive intensity-modulated radiotherapy (IMRT) of 70 Gy will be given in 33 fractions.
  Other Names:
  IMRT
  Arms: Induction GP+placebo group

SUMMARY:
The main questions it aims to answer are:

1. Does the combination of GP induction chemotherapy and toripalimab improve the 3-year progression-free survival (PFS) compared to GP induction chemotherapy with placebo?
2. What are the differences in CR after induction therapy, 3-year overall survival (OS), locoregional progression, and distant progression between the two groups?
3. What are the differences in safety between the two groups?
4. Are there predictive biomarkers of therapeutic efficacy, such as changes in EBV DNA or immune parameters, that correlate with treatment outcomes?

Researchers will compare the GP + toripalimab group with the GP + placebo group to see if the toripalimab combination shows superior efficacy.

Participants will:

Receive either GP chemotherapy with toripalimab or GP chemotherapy with placebo as induction therapy.

Undergo concurrent chemoradiotherapy ± adjuvant metronomic capecitabine following induction therapy.

Be monitored closely for safety and efficacy outcomes.

DETAILED DESCRIPTION:
Platinum-based concurrent chemoradiotherapy is the standard of care for patients with locoregionally advanced nasopharyngeal carcinoma (NPC). Gemcitabine plus cisplatin (GP) has been demonstrated an effective chemotherapy regimen for NPC patients in previous studies. The results of GP combined with concurrent chemoradiotherapy in the treatment of locoregionally advanced nasopharyngeal carcinoma showed 10% of locoregionally advanced NPC patients had complete response after three cycles of GP induction chemotherapy, and GP induction chemotherapy added to chemoradiotherapy significantly improved recurrence-free survival (85.3% vs 76.5%) and overall survival (94.6% vs 90.3%) among locoregionally advanced NPC patients , as compared with chemoradiotherapy alone. Therefore, GP regimen has been established as the highest level of evidence-based induction chemotherapy in the 2020 National Comprehensive Cancer Network (NCCN) guidelines. Despite this intensified treatment approach, 20-30% of patients still have disease recurrences, highlighting the need for novel treatments in this population. Anti-PD-1 therapy and chemotherapy is a recommended first-line treatment for recurrent or metastatic nasopharyngeal carcinoma. So we hypothesize that GP induction chemotherapy combined with toripalimab could further improve survival of patients with locoregionally advanced NPC. The goal of this randomized, double-blind, controlled phase III clinical trial is to evaluate the efficacy and safety of the GP induction chemotherapy combined with toripalimab or placebo , followed by concurrent chemoradiotherapy ± adjuvant metronomic capecitabine in patients with high-risk locoregionally advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participates and signs an informed consent form.
2. Aged 18-70 years, male or non-pregnant female.
3. Pathologically confirmed nasopharyngeal non-keratinizing carcinoma (differentiated or undifferentiated, i.e., WHO Type II or III).
4. Staging of any T, N2-3 or T4N1 (9th AJCC/UICC staging), with no distant metastasis.
5. ECOG performance status score of 0-1.
6. Hemoglobin (HGB) ≥90 g/L, neutrocyte count≥1.5×10⁹/L, platelets (PLT) ≥100×10⁹ /L.
7. Liver function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤2.5×upper limit of normal (ULN), and bilirubin ≤ 1.5×ULN.
8. Adequate renal function: creatinine clearance rate ≥ 60 ml/min (Cockcroft-Gault formula).
9. Women of childbearing potential (WOCBP) who are sexually active must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of the study drug. Men who are sexually active with WOCBP must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of the study drug.

Exclusion Criteria:

1. Age > 70 years or < 18 years.
2. Patients with recurrence or distant metastases.
3. Pathologically confirmed nasopharyngeal keratinizing squamous cell carcinoma (WHO Type I).
4. Patients who have previously undergone radiotherapy or systemic chemotherapy.
5. Hepatitis B surface antigen (HBsAg) positive and hepatitis B virus DNA >1000 copies/ml or 200IU/ml.
6. Hepatitis C virus (HCV) antibody positive.
7. Has active autoimmune disease, except type I diabetes, hypothyroidism treated with replacement therapy, and skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia).
8. Has any condition that required systemic corticosteroid (equivalent to prednisone >10mg/d) or other immunosuppressive therapy within 28 days before informed consent. Patients who received systemic corticosteroid equivalent to prednisone ≤10mg/d, inhale or topical corticosteroids will be allowed.
9. Has a known history of active bacillus tuberculosis within 1 year; patients with adequately treated active bacillus tuberculosis over 1 year ago will be allowed.
10. Has a known history of interstitial lung disease.
11. Has received a live vaccine within 30 days before informed consent or will receive a live vaccine in the near future.
12. Is pregnant or breastfeeding.
13. Prior malignancy within 5 years, except in situ cancer, adequately treated non-melanoma skin cancer and papillary thyroid carcinoma.
14. Has known allergy to large molecule protein products or any compound of toripalimab.
15. Has a known history of human immunodeficiency virus infection.
16. Any other condition, including symptomatic heart failure, unstable angina, myocardial infarction, active infection requiring systemic therapy, mental illness, or domestic/social factors, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study or interferes with the interpretation of the results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 3 years
  Defined as the time from randomisation to first progression (locoregional or distant) or death, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival | 3 years
  Defined as the time from randomization to death from any cause.
Locoregional Progression | 3 years
  Defined as the time from randomization to the occurrence of a locoregional progression. Cumulative incidence of locoregional progression will be calculated within a competing risk framework (Fine and Gray 1999).
Distant Progression | 3 years
  Defined as the time from randomization to the occurrence of a distant progression. Cumulative incidence of distant progression will be calculated within a competing risk framework (Fine and Gray 1999).
Complete Response Rate | 9 weeks
  CR assessed by investigator, according to the Response Evaluation Criteria in Solid Tumors (RECIST1.1) from the National Cancer Institute (NCI). Disease response evaluated after the completion of the induction therapy. Complete response defined as the complete disappearance of the target and non-target lesion(s) identified at baseline after radiological evaluation by Magnetic Resonance Imaging (MRI) .
Incidence of Acute and Late Toxicity | 3 years
  Incidence of acute toxicity is calculated for each adverse event respectively and severity is evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE) 5.0 criteria. Late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme.

OTHER OUTCOMES:
The correlation of pre-treatement plasma EBV DNA and dynamic change after induction therapy between with the PFS | 3 years
  Plasma EBV DNA testing will be conducted before treatment and after induction therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mai HQ, Chen QY, Chen D, Hu C, Yang K, Wen J, Li J, Shi YR, Jin F, Xu R, Pan J, Qu S, Li P, Hu C, Liu YC, Jiang Y, He X, Wang HM, Lim WT, Liao W, He X, Chen X, Liu Z, Yuan X, Li Q, Lin X, Jing S, Chen Y, Lu Y, Hsieh CY, Yang MH, Yen CJ, Samol J, Feng H, Yao S, Keegan P, Xu RH. Toripalimab or placebo plus chemotherapy as first-line treatment in advanced nasopharyngeal carcinoma: a multicenter randomized phase 3 trial. Nat Med. 2021 Sep;27(9):1536-1543. doi: 10.1038/s41591-021-01444-0. Epub 2021 Aug 2. PMID 34341578
- [Background] Chen YP, Liu X, Zhou Q, Yang KY, Jin F, Zhu XD, Shi M, Hu GQ, Hu WH, Sun Y, Wu HF, Wu H, Lin Q, Wang H, Tian Y, Zhang N, Wang XC, Shen LF, Liu ZZ, Huang J, Luo XL, Li L, Zang J, Mei Q, Zheng BM, Yue D, Xu J, Wu SG, Shi YX, Mao YP, Chen L, Li WF, Zhou GQ, Sun R, Guo R, Zhang Y, Xu C, Lv JW, Guo Y, Feng HX, Tang LL, Xie FY, Sun Y, Ma J. Metronomic capecitabine as adjuvant therapy in locoregionally advanced nasopharyngeal carcinoma: a multicentre, open-label, parallel-group, randomised, controlled, phase 3 trial. Lancet. 2021 Jul 24;398(10297):303-313. doi: 10.1016/S0140-6736(21)01123-5. Epub 2021 Jun 7. PMID 34111416
- [Background] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593